CLINICAL TRIAL: NCT00314834
Title: Effect of Intradialytic Parenteral Nutrition on Morbidity and Mortality of Malnourished Hemodialysis Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: EZUS-LYON 1 (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Societe Francaise de Dialyse (Unknown); Societe Francophone de Nutrition Enterale et Parenterale (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZUS-A1244
Record Dates: First submitted 2006-04-14; First posted 2006-04-17 (Estimated); Last update posted 2006-04-17 (Estimated); Status verified 2005-03

CONDITIONS: Hemodialysis; Malnutrition
Keywords: hemodialysis; intradialytic parenteral nutrition; oral supplementation; survival; hospitalization; serum albumin; prealbumin; transthyretin
MeSH Terms: conditions — Malnutrition

INTERVENTIONS:
Drug: Intradialytic parenteral nutrition

SUMMARY:
IDPN is widely used in HD patients without clue of its effectiveness. Study objectives: to evaluate IDPN effects on mortality (main objective), hospitalization rates, nutritional status, dialysis efficacy, Karnofsky score

DETAILED DESCRIPTION:
IDPN is widely used in HD patients without clue of its effectiveness. Study objectives: to evaluate IDPN effects on mortality (main objective), hospitalization rates, nutritional status, dialysis efficacy, Karnofsky score.

Patient eligibility: adult patients ≤ 82 y with HD vintage > 6 mo. and 2 of the following malnutrition criteria: BMI ≤ 20 kg/m2, BW loss/6 mo. ≥ 10%, serum albumin ≤ 35 g/L, prealbumin ≤ 300 mg/L.

Recruitment: patients in 38 HD units from January 2001 to December 2002 Study protocol. Patients are randomized into 2 groups: IDPN group, given IDPN during one year, and control group. For ethical reasons, the 2 groups are given oral supplementation during the same period.

Follow-up: two years after start of nutritional therapy. Study end: December 31, 2004. Final results will be available in early 2005.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 82 years
* hemodialysis vintage more than 6 months
* two of the following markers of malnutrition:
* body mass index (BMI) <= 20 kg/m2
* body weight loss within 6 months >= 10 percent
* serum albumin <= 35 g/L
* prealbumin <= 300 mg/L

Exclusion Criteria:

* weekly dialysis time < 12 h
* urea Kt/V index < 1.2
* serum albumin > 38 g/L
* prealbumin > 330 mg/L
* hypertriglyceridemia > 2.5 mmol/L
* associated comorbidities compromising the one-year survival
* treatment by oral, enteral or parenteral feeding during the last 3 months
* hospitalization at time of randomization

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204
Dates: Start 2001-01; Study Completion 2004-12

PRIMARY OUTCOMES:
mortality

SECONDARY OUTCOMES:
hospitalization rate, Karnofsky score, BMI, serum albumin and prealbumin

CONTACTS AND LOCATIONS:
Overall Officials: Noel JM Cano, MD-PhD, Study Director

REFERENCES:
- [Derived] Cano NJ, Fouque D, Roth H, Aparicio M, Azar R, Canaud B, Chauveau P, Combe C, Laville M, Leverve XM; French Study Group for Nutrition in Dialysis. Intradialytic parenteral nutrition does not improve survival in malnourished hemodialysis patients: a 2-year multicenter, prospective, randomized study. J Am Soc Nephrol. 2007 Sep;18(9):2583-91. doi: 10.1681/ASN.2007020184. Epub 2007 Jul 26. PMID 17656473